CLINICAL TRIAL: NCT01245062
Title: A Phase III Randomized, Open-label Study Comparing GSK1120212 to Chemotherapy in Subjects With Advanced or Metastatic BRAF V600E/K Mutation-positive Melanoma
Brief Title: GSK1120212 vs Chemotherapy in Advanced or Metastatic BRAF V600E/K Mutation-positive Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114267
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-01

CONDITIONS: Melanoma
Keywords: MEK inhibitor; Cancer; Metastatic Melanoma; BRAF mutant metastatic melanoma; GSK1120212
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — trametinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GSK1120212 (Experimental): MEK inhibitor
  Interventions: Drug: GSK1120212
- Chemotherapy (Active Comparator): Investigator Choice of DTIC or paclitaxel
  Interventions: Drug: Chemotherapy
- Crossover (Experimental): MEK inhibitor after documented progression on Chemotherapy Arm
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — MEK inhibitor
  Arms: Crossover; GSK1120212
Drug: Chemotherapy — Investigator Choice of DTIC or paclitaxel
  Arms: Chemotherapy

SUMMARY:
This is a two-arm, open-label, randomized Phase III study comparing single agent GSK1120212 to chemotherapy (either dacarbazine or paclitaxel) in subjects with Stage IIIc or Stage IV malignant cutaneous melanoma. All subjects must have a BRAF mutation-positive tumour sample. Subjects who have received up to one prior regimen of chemotherapy in the advanced or metastatic melanoma setting will be enrolled into the study. Subjects with any prior BRAF or MEK inhibitor use will be excluded. Approximately 297 subjects will be enrolled with 2:1 randomization (198 subjects into the GSK1120212 arm and 99 subjects into the chemotherapy arm). The primary endpoint for the statistical analysis will be a comparison of progression free survival for subjects receiving GSK1120212 compared to chemotherapy. Subjects who have progression on chemotherapy will be offered the option to receive GSK1120212.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Stage III unresectable (Stage IIIc) or metastatic (Stage IV) cutaneous melanoma which is also determined to be BRAF V600E/K mutation-positive by the central laboratory
* Received no prior treatment or up to one prior regimen of chemotherapy for advanced or metastatic melanoma. Prior treatment with immunotherapy (with the exception of prior ipilimumab, which is only allowed if given in the adjuvant setting), cytokine therapy, biological or vaccine regimen is permitted. Prior use of sorafenib is allowed
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Women of childbearing potential and men with reproductive potential must agree to use effective contraception during the study. Additionally women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate screening organ function

Exclusion Criteria:

* Any prior use of BRAF inhibitors or MEK inhibitors.
* Subjects who have received dacarbazine or paclitaxel prior to randomization will not be eligible to receive the same chemotherapy as study medication (i.e. a subject who received prior dacarbazine cannot receive dacarbazine on this trial and would thus receive paclitaxel if randomized to the control arm)
* History of another malignancy. Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled. Consult GSK Medical Monitor if unsure whether second malignancies meet requirements specified above
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which will be allowed)
* Brain metastases with the following exceptions that are ALL confirmed by the GSK Medical Monitor:

All known lesions must be previously treated with surgery or stereotactic radiosurgery, and Brain lesion(s), if still present, must be confirmed stable (i.e. no increase in lesion size) for ≥90 days prior to randomization (must be documented with two consecutive MRI or CT scans using contrast), and asymptomatic with no corticosteroids requirement for ≥ 30 days prior to randomization, and no enzyme-inducing anticonvulsants for ≥ 30 days prior to randomization

* History or evidence of cardiovascular risk including any of the following:

  * QTcB ≥ 480 msec.
  * History or evidence of current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation for >30 days prior to randomization are eligible
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization.
  * History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association
* History of interstitial lung disease or pneumonitis
* History or current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR):

  * History of RVO or CSR, or predisposing factors to RVO or CSR (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes).
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:
* Evidence of new optic disc cupping.
* Intraocular pressure > 21 mm Hg as measured by tonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2011-10-26 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (105):
- United States (13):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
- GSK Investigational Site, Buenos Aires, Argentina
- Australia (10):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Port Macquarie, New South Wales
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Townsville, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Kurralta Park, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Austria (2):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Vienna
- Belgium (8):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Jette
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk
  - GSK Investigational Site, Yvoir
- Canada (9):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Czechia (4):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Zlín
- France (9):
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Villejuif
- Germany (10):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Buxtehude, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
- New Zealand (3):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Newtown, Wellington
- GSK Investigational Site, Oslo, Norway
- Poland (2):
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Russia (4):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Magnitogorsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- GSK Investigational Site, Zurich, Switzerland
- Ukraine (8):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Sumy
  - GSK Investigational Site, Sympheropol
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Uzhhorod
- United Kingdom (11):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Southampton

REFERENCES:
- [Background] KT Flaherty, C Robert, P Hersey, P Nathan, C Garbe, M Milhem, L Demidov, J Hassel, P Rutkowski, P Mohr, R Dummer, U Trefzer, JMG Larkin, J Utikal, B Dreno, M Nyakas, MR Middleton, JC Becker, M Casey, LJ Sherman, FS Wu, D Ouellet, AM Martin, K Patel, & D S. MEK inhibition improves survival in Melanoma with activating BRAF Mutations. [N Engl J Med]. 2012;367:107-14.
- [Result] Flaherty KT, Robert C, Hersey P, Nathan P, Garbe C, Milhem M, Demidov LV, Hassel JC, Rutkowski P, Mohr P, Dummer R, Trefzer U, Larkin JM, Utikal J, Dreno B, Nyakas M, Middleton MR, Becker JC, Casey M, Sherman LJ, Wu FS, Ouellet D, Martin AM, Patel K, Schadendorf D; METRIC Study Group. Improved survival with MEK inhibition in BRAF-mutated melanoma. N Engl J Med. 2012 Jul 12;367(2):107-14. doi: 10.1056/NEJMoa1203421. Epub 2012 Jun 4. PMID 22663011
- [Derived] Robert C, Flaherty K, Nathan P, Hersey P, Garbe C, Milhem M, Demidov L, Mohr P, Hassel JC, Rutkowski P, Dummer R, Utikal J, Kiecker F, Larkin J, D'Amelio A Jr, Mookerjee B, Schadendorf D. Five-year outcomes from a phase 3 METRIC study in patients with BRAF V600 E/K-mutant advanced or metastatic melanoma. Eur J Cancer. 2019 Mar;109:61-69. doi: 10.1016/j.ejca.2018.12.015. Epub 2019 Jan 25. PMID 30690294
- [Derived] Latimer NR, Bell H, Abrams KR, Amonkar MM, Casey M. Adjusting for treatment switching in the METRIC study shows further improved overall survival with trametinib compared with chemotherapy. Cancer Med. 2016 May;5(5):806-15. doi: 10.1002/cam4.643. Epub 2016 Jan 27. PMID 27172483
- [Derived] Santiago-Walker A, Gagnon R, Mazumdar J, Casey M, Long GV, Schadendorf D, Flaherty K, Kefford R, Hauschild A, Hwu P, Haney P, O'Hagan A, Carver J, Goodman V, Legos J, Martin AM. Correlation of BRAF Mutation Status in Circulating-Free DNA and Tumor and Association with Clinical Outcome across Four BRAFi and MEKi Clinical Trials. Clin Cancer Res. 2016 Feb 1;22(3):567-74. doi: 10.1158/1078-0432.CCR-15-0321. Epub 2015 Oct 7. PMID 26446943
- [Derived] Schadendorf D, Amonkar MM, Milhem M, Grotzinger K, Demidov LV, Rutkowski P, Garbe C, Dummer R, Hassel JC, Wolter P, Mohr P, Trefzer U, Lefeuvre-Plesse C, Rutten A, Steven N, Ullenhag G, Sherman L, Wu FS, Patel K, Casey M, Robert C. Functional and symptom impact of trametinib versus chemotherapy in BRAF V600E advanced or metastatic melanoma: quality-of-life analyses of the METRIC study. Ann Oncol. 2014 Mar;25(3):700-706. doi: 10.1093/annonc/mdt580. Epub 2014 Feb 6. PMID 24504441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized open-label, multi-center Phase III study to evaluate the efficacy and safety of single agent trametinib compared with chemotherapy (CT) (dacarbazine or paclitaxel). Participants (par.) were enrolled by 86 sites in 19 countries from December 2010 to July 2011. Results as of 16 December 2016 data-cut have been presented.
Pre-assignment Details: Participants (par.) were stratified for lactate dehydrogenase and prior CT for advanced or metastatic disease. 1059 par. were screened and 322 were enrolled to receive trametinib (214 par.) or CT (108 par.) until disease progression, death, or withdrawal. Par. randomized to CT were allowed to cross-over to trametinib if disease progressed.
Groups:
- Trametinib: Participants with histologically confirmed cutaneous advanced or metastatic melanoma (Stage IIIC or Stage IV), with a BRAF (a human gene encoding for protein called B-Raf, which is involved in a signaling pathway and is important for cell growth) V600 E/K mutation-positive tumor sample as determined via the central BRAF mutation assay, received a Trametinib 2 milligram (mg) tablet once daily until disease progression, death, or withdrawal.
- Chemotherapy: Participants with histologically confirmed cutaneous advanced or metastatic melanoma (Stage IIIC or Stage IV), with a BRAF V600 E/K mutation-positive tumor sample as determined via the central BRAF mutation assay, received an intravenous (IV) dose of Dacarbazine 1000 mg per square meter every 3 weeks or Paclitaxel 175 mg per square meter every 3 weeks at the discretion of the investigator, provided the participant had not received that type of chemotherapy before randomization, until disease progression, death, or withdrawal.
- Cross-over From Chemotherapy to Trametinib: Participants randomized to chemotherapy and who did not receive subsequent anti-cancer therapy after discontinuing chemotherapy were allowed to cross-over to Trametinib and received 2 mg tablet once daily until disease progression, death or withdrawal.
Period: Randomization and Crossover Phase
Arm/Group | Trametinib | Chemotherapy | Cross-over From Chemotherapy to Trametinib
Started (Par. randomized onto study.) | 214 | 108 | 0
Completed (Par. completed the study as they died during the conduct of the study.) | 173 | 77 | 0
Not Completed | 41 | 31 | 0
Not completed — Lost to Follow-up | 4 | 2 | 0
Not completed — Physician Decision | 2 | 4 | 0
Not completed — Withdrew Consent | 12 | 11 | 0
Not completed — Study closed/ terminated | 23 | 14 | 0
Period: Cross-over Phase
Arm/Group | Trametinib | Chemotherapy | Cross-over From Chemotherapy to Trametinib
Started | 0 | 0 | 70 (As of the data cut on December 16, 2016, 70 of 108 participants crossed over from CT to trametinib.)
Completed (Par. completed the study as they died during the conduct of the study.) | 0 | 0 | 53
Not Completed | 0 | 0 | 17
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrew Consent | 0 | 0 | 4
Not completed — Study closed/ terminated | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trametinib | Chemotherapy | Total
Number analyzed (Participants) | 214 | 108 | 322
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (12.97) | 52.8 (13.56) | 53.8 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 55 | 149
  Male | 120 | 53 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: White - Arabic/North African Heritage | 2 | 0 | 2
  Race/Ethnicity, Customized: White - White/Caucasian/European Heritage | 212 | 107 | 319
  Race/Ethnicity, Customized: White - Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival in BRAF V600E Mutation-positive Participants Without a History of Brain Metastases as Assessed by the Investigator and Independent Review
Description: Progression-free survival (PFS) is defined as the time from randomization to the first documented occurrence of disease progression (PD) or death. PFS for investigator-assessed and blinded, independent, central review committee (BRIC)-assessed responses was summarized per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1, which is a set of published rules defining when cancer participants improve (respond), stay the same (stabilize), or worsen (progress) during treatment. Disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of at least 1 new lesion, or the worsening of non-target lesions significant enough to require study treatment discontinuation. Primary Efficacy Population included all participants with BRAF V600E mutation-positive melanoma without a history of brain metastases.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 178 | 95
Months
  Investigator-Assessed | 4.8 [3.5 to 4.9] | 1.4 [1.4 to 2.7]
  Independent Review | 4.9 [4.5 to 5.1] | 1.6 [1.4 to 2.8]
Statistical Analysis 1: Comparison: Trametinib vs Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank — P-value from a stratified log-rank test was adjusted for prior chemotherapy for advanced or metastatic disease and Baseline lactate dehydrogenase; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.31 to 0.64] — Investigator-Assessed PFS. HR <1 indicates a lower risk with Trametinib compared with CT. HR from a stratified log-rank test was adjusted for prior chemotherapy for advanced or metastatic disease and Baseline lactate dehydrogenase
Statistical Analysis 2: Comparison: Trametinib vs Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.29 to 0.60] — Independent Review PFS. HR <1 indicates a lower risk with Trametinib compared with CT. HR from a stratified log-rank test was adjusted for prior chemotherapy for advanced or metastatic disease and Baseline lactate dehydrogenase

2. Secondary Outcome: Progression-free Survival in All Participants
Description: PFS is defined as the time from the date of randomization to the first documented occurrence of PD or death. Investigator-assessed and BRIC-assessed PFS were summarized per RECIST, Version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation. Intend-To-Treat (ITT) Population included all randomized participants regardless of whether or not treatment was administered.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 214 | 108
Months
  Investigator-Assessed | 4.9 [4.5 to 5.0] | 1.5 [1.4 to 2.8]
  Independent radiologist assessed-Assessed | 4.9 [4.6 to 5.0] | 1.5 [1.4 to 2.8]

3. Secondary Outcome: PFS in BRAF V600E Mutation-positive Participants Without a History of Brain Metastases and Without Prior Chemotherapy as Assessed by the Investigator
Description: PFS is defined as the time from the date of randomization to the first documented occurrence of PD or death. Investigator-assessed PFS was summarized per RECIST, Version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 114 | 62
Months | 4.8 [3.4 to 5.0] | 1.4 [1.4 to 1.7]

4. Secondary Outcome: PFS in BRAF V600E Mutation-positive Participants Without a History of Brain Metastases and With Prior Chemotherapy as Assessed by the Investigator
Description: as for outcome 3
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 64 | 33
Months | 4.8 [2.9 to 4.9] | 2.7 [1.4 to 2.9]

5. Secondary Outcome: Overall Survival in All Participants
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: Day 1 until death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 214 | 108
Months | 15.6 [13.5 to 17.3] | 11.3 [7.2 to 14.8]

6. Secondary Outcome: Overall Survival in BRAF V600E Mutation-positive Participants Without a History of Brain Metastases
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause. NA indicates data was not available.
Time Frame: Day 1 until death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 178 | 95
Months | NA [NA to NA] — At the time of this report, there was limited follow-up for survival; therefore, the median and the confidence interval (CI) could not be estimated. | NA [6.8 to NA] — At the time of this report, there was limited follow-up for survival; therefore, the median and the upper limit (UL) of the CI could not be estimated.

7. Secondary Outcome: Number of BRAF V600E Mutation-positive Participants Without a History of Brain Metastases With Overall Response (OR) as Assessed by the Investigator and Independent Review
Description: OR is defined as the number of participants with evidence of complete response (CR; disappearance of all target lesions. Any pathological lymph node must be less than 10 mm in the short axis) or partial response (PR: at least a 30% decrease in the sum of the diameters of target lesions) evaluated by the Investigator and an independent review per RECIST, Version 1.1.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Number; unit: Participants
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 178 | 95
Participants
  Investigator-Assessed: CR | 4 | 0
  Investigator-Assessed: PR | 39 | 7
  Independent Review: CR | 0 | 0
  Independent Review: PR | 33 | 3

8. Secondary Outcome: Number of Participants With OR as Assessed by the Investigator and Independent Review
Description: OR is defined as the number of participants with evidence of complete response (disappearance of all target lesions. Any pathological lymph node must be less than 10 mm in the short axis) or partial response (at least a 30% decrease in the sum of the diameters of target lesions) evaluated by the Investigator and an independent review per RECIST, Version 1.1.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 214 | 108
Participants
  Investigator-Assessed: CR | 8 | 2
  Investigator-Assessed: PR | 53 | 8
  Independent Review: CR | 0 | 1
  Independent Review: PR | 41 | 4

9. Secondary Outcome: Number of BRAF V600E Mutation-positive Participants Classified as Confirmed Responders (CR and PR) as Assessed by the Investigator
Description: OR is defined as the number of participants with evidence of complete response (disappearance of all extranodal lesions. Any pathological lymph node must be less than 10 mm in the short axis) or partial response (at least a 30% decrease in the sum of the diameters of target lesions) evaluated by the Investigator per RECIST, Version 1.1.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 184 | 97
Participants
  V600E Mutation, CR | 4 | 0
  V600E Mutation, PR | 40 | 7

10. Secondary Outcome: Number of BRAF V600K Mutation-positive Participants Classified as Confirmed Responders (CR and PR) as Assessed by the Investigator
Description: OR is defined as the number of participants with evidence of complete response (CR; disappearance of all extranodal lesions. Any pathological lymph node must be less than 10 mm in the short axis) or partial response (PR: at least a 30% decrease in the sum of the diameters of target lesions) evaluated by the Investigator per RECIST, Version 1.1.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 29 | 11
Participants
  V600K Mutation, CR | 0 | 0
  V600K Mutation, PR | 3 | 2

11. Secondary Outcome: Number of Participants With OR Following Cross-over to Trametinib
Description: OR is defined as the number of participants with evidence of CR (disappearance of all target lesions. Any pathological lymph node must be less than 10 millimeters in the short axis) or PR (at least a 30% decrease in the sum of the diameters of target lesions) evaluated by the Investigator in participants following cross-over to Trametinib. The evaluation was carried out by the Investigator per RECIST, Version 1.1. Cross-over Population included the subset of participants who were randomized to CT and who elected to cross-over to Trametinib following disease progression on CT. Only participants who received at least one dose of Trametinib were included in this population.
Time Frame: Day 1 of cross-over therapy until the earliest date of disease progression or death due to any cause (average of 18.3 months)
Population: Cross-over Population
Measure: Number; unit: Participants
Arm/Group | Cross-over From Chemotherapy to Trametinib
Number analyzed (Participants) | 70
Participants
  CR | 2
  PR | 29

12. Secondary Outcome: Duration of Response (DoR) for All BRAF V600E Mutation-positive Participants Without a Prior History of Brain Metastases Classified as Confirmed Responders (CR or PR) as Assessed by the Investigator Review
Description: DoR is defined as the time from the first documented evidence of CR (disappearance of all target lesions. Any pathological lymph node must be less than 10 mm in the short axis) or PR (at least a 30% decrease in the sum of the diameters of target lesions) until PD (at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation) or death due to any cause. DoR for the investigator-assessed (INVA) response data were summarized per RECIST, Version 1.1. Only those participants with confirmed response (CR and PR) were analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 43 | 7
Months | 5.5 [4.9 to 5.9] | NA [3.5 to NA] — There were too few events to provide an estimable median or UL of the CI.

13. Secondary Outcome: DoR for All BRAF V600E Mutation-positive Participants Without a Prior History of Brain Metastases Classified as Confirmed Responders (CR or PR) as Assessed by the Independent Review
Description: DoR is defined as the time from the first documented evidence of CR (disappearance of all target lesions. Any pathological lymph node must be less than 10 mm in the short axis) or PR (at least a 30% decrease in the sum of the diameters of target lesions) until PD (at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation) or death due to any cause. DoR for the independently-assessed (INDA) response data were summarized per RECIST, Version 1.1. Only those participants with confirmed response (CR and PR) were analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 33 | 3
Months | 5.6 [3.8 to 5.9] | NA [3.5 to NA] — There were too few events to provide an estimable median or UL of the CI.

14. Secondary Outcome: DoR for All Confirmed Responders (CR or PR) as Assessed by the Investigator Review
Description: DoR is defined as the time from the first documented evidence of CR (disappearance of all target lesions. Any pathological lymph node must be less than 10 mm in the short axis) or PR (at least a 30% decrease in the sum of the diameters of target lesions) until PD or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation. DoR for the INVA response data was summarized per RECIST, Version 1.1. Only those participants with confirmed response (CR and PR) were analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 47 | 9
Months | 5.5 [4.1 to 5.9] | NA [5.0 to NA] — There were too few events to provide an estimable median or UL of the CI.

15. Secondary Outcome: DoR for All Confirmed Responders (CR or PR) as Assessed by the Independent Review
Description: DoR is defined as the time from the first documented evidence of CR (disappearance of all target lesions. Any pathological lymph node must be less than 10 mm in the short axis) or PR (at least a 30% decrease in the sum of the diameters of target lesions) until PD or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation. DoR for the INDA response data was summarized per RECIST, Version 1.1. Only those participants with confirmed response (CR and PR) were analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: Day 1 until the earliest date of disease progression or death due to any cause (average of 20.3 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib | Chemotherapy
Number analyzed (Participants) | 41 | 5
Months | 5.6 [4.1 to 5.9] | NA [5.0 to NA] — There were too few events to provide an estimable median or UL of the CI.

16. Secondary Outcome: DoR for All Responders (CR or PR) Following Cross-over to Trametinib as Assessed by the Investigator
Description: DoR is defined as the time from the first documented evidence of CR (disappearance of all extra nodal lesions. Any pathological lymph node must be less than 10 mm in the short axis) or PR (at least a 30% decrease in the sum of the diameters of target lesions) until PD or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation. DoR data were summarized per RECIST, Version 1.1Only those participants with confirmed response (CR and PR) were analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data was not available.
Time Frame: as for outcome 11
Population: Cross-over Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cross-over From Chemotherapy to Trametinib
Number analyzed (Participants) | 13
Months | 2.7 [1.3 to NA] — There were too few events to provide an estimable UL of the CI.

17. Secondary Outcome: PFS Following Cross-over to Trametinib as Assessed by the Investigator
Description: PFS is defined as the time from the first dose of cross-over therapy to the first documented occurrence of PD or death. PFS was summarized per RECIST, Version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation.
Time Frame: as for outcome 11
Population: Cross-over Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cross-over From Chemotherapy to Trametinib
Number analyzed (Participants) | 70
Months | 3.0 [2.7 to 4.8]

ADVERSE EVENTS:
Time Frame: Participants were analyzed from the first dose of study medication to 28 days after discontinuation of study medication (average of 20.3 months in the Randomization Phase and 18.3 months in the Cross-over Phase).
Description: Serious adverse events (SAEs) and non-serious AEs were collected in the Safety Population, comprised of all randomized participants included in the study who received at least one dose of study medication.
Arm/Group | Trametinib | Chemotherapy | Cross-over From Chemotherapy to Trametinib
All-Cause Mortality (participants affected / at risk) | 172/211 | 22/99 | 53/70
Serious Adverse Events (participants affected / at risk) | 52/211 | 19/99 | 18/70
Other Adverse Events (participants affected / at risk) | 207/211 | 88/99 | 66/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib (N=211) | Chemotherapy (N=99) | Cross-over From Chemotherapy to Trametinib (N=70)
Cellulitis (Infections and infestations) | 4 | 0 | 2
Erysipelas (Infections and infestations) | 5 | 0 | 1
Infection (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Localized infection (Infections and infestations) | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 4 | 2
Axillary pain (General disorders) | 0 | 1 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0
Edema (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Hemoglobin decreased (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Corneal graft rejection (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Ischemic stroke (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Infected seroma (Infections and infestations) | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib (N=211) | Chemotherapy (N=99) | Cross-over From Chemotherapy to Trametinib (N=70)
Rash (Skin and subcutaneous tissue disorders) | 123 | 10 | 37
Alopecia (Skin and subcutaneous tissue disorders) | 38 | 19 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 42 | 2 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 1 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 1 | 10
Eczema (Skin and subcutaneous tissue disorders) | 12 | 0 | 6
Diarrhea (Gastrointestinal disorders) | 94 | 16 | 24
Nausea (Gastrointestinal disorders) | 48 | 39 | 12
Constipation (Gastrointestinal disorders) | 34 | 22 | 12
Vomiting (Gastrointestinal disorders) | 33 | 21 | 16
Dry mouth (Gastrointestinal disorders) | 19 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 19 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 16 | 3 | 4
Stomatitis (Gastrointestinal disorders) | 13 | 1 | 0
Fatigue (General disorders) | 62 | 29 | 8
Asthenia (General disorders) | 12 | 12 | 4
Pyrexia (General disorders) | 15 | 8 | 6
Mucosal inflammation (General disorders) | 15 | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 10 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 9 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 8 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0
Headache (Nervous system disorders) | 30 | 15 | 0
Paraesthesia (Nervous system disorders) | 10 | 9 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 9 | 0
Hypertension (Vascular disorders) | 40 | 9 | 9
Lymphedema (Vascular disorders) | 18 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 6 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 1 | 4
Folliculitis (Infections and infestations) | 22 | 2 | 6
Paronychia (Infections and infestations) | 26 | 1 | 10
Aspartate aminotransferase increased (Investigations) | 21 | 1 | 7
Alanine aminotransferase increased (Investigations) | 16 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 13 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 5 | 0
Platelet count decreased (Investigations) | 1 | 5 | 0
Anemia (Blood and lymphatic system disorders) | 13 | 10 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 18 | 10 | 6
Insomnia (Psychiatric disorders) | 15 | 7 | 4
Oedema peripheral (General disorders) | 55 | 2 | 16
Nasopharyngitis (Infections and infestations) | 15 | 4 | 0
Rash pustular (Infections and infestations) | 11 | 0 | 5
Dysgeusia (Nervous system disorders) | 12 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 6 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 21 | 0 | 9
Inflammation (General disorders) | 0 | 0 | 4
Influenza like illness (General disorders) | 0 | 0 | 4
Peripheral swelling (General disorders) | 0 | 0 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 4
Nail infection (Infections and infestations) | 0 | 0 | 4
Weight decreased (Investigations) | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 7
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.